CLINICAL TRIAL: NCT05853419
Title: Change History and Adopt a Robotic SolutioN for anGioplasty procedurE
Acronym: CHANGE
Status: Recruiting | Type: Observational
Sponsor: Robocath (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: ROB-03
Record Dates: First submitted 2023-02-28; First posted 2023-05-10 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population: Adult patients with coronary artery disease and a clinical indication for PCI
  Interventions: Device: Robotic-assisted PCI

INTERVENTIONS:
Device: Robotic-assisted PCI — Robotic-assisted PCI will be performed according to the routine hospital practices, current scientific guidelines and following Instructions for Use (IFU) provided by the manufacturer

SUMMARY:
The main objective of the CHANGE registry is the evaluation of the real-world performance and safety profile of the R-One System in PCI.

DETAILED DESCRIPTION:
The R-One system is a class "IIb" CE marked medical device designed to remote deliver and manipulate coronary guidewires and stent/balloon devices during Percutaneous Coronary Intervention (PCI). The system comprises the R-One Robotic Platform used in combination with two accessories, the Mobile Radioprotection Screen and a sterile and single-use R-One Consumable Kit. The R-One is not autonomous and operates only under the operator's commands.

This study is a single-arm, open-label, multi-center registry.

The CHANGE registry, part of the ROBOCATH's post-market clinical follow-up activities, is a real world study aiming to confirm the safety and performance, including the clinical benefit, of the R-One robotic systems medical device.

500 patients with coronary artery disease and with clinical indication for PCI will be recruited in up to Up to 15 centers distributed in Europe and South Africa.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years;
* 2.Subjects with coronary artery disease with clinical indication for PCI;
* 3.Subject deemed appropriate for robotic-assisted PCI; and
* 4.The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

* 1.Failure/inability/unwillingness to provide informed consent, unless the ethic committee has waived informed consent; or
* 2.The Investigator determines that the subject or the coronary anatomy is not suitable for robotic-assisted PCI.
* 3.STEMI
* 4.Cardiogenic shock
* 5.Subjects will not be included if they are under judicial protection, guardianship or curatorship or if they are deprived of their liberty by judicial or administrative decision.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease and a clinical indication for PCI
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical success | From Day 0 to Day 3
  Less than 30% residual stenosis (visual estimate) post PCI in the lesion(s) treated with the R-One System, without in-hospital major adverse cardiac events (MACE).
Technical success | During procedure
  Absence of any unplanned manual assistance or conversion to manual PCI for procedural completion

SECONDARY OUTCOMES:
Radiation exposure for the patient | During procedure
  Dose (DSP and Air Kerma) measured by the imaging system during the procedure.
Overall Procedure Time | During procedure
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
Overall contrast volume | During procedure
  Total volume of contrast (mL) used during the procedure.
Radiation exposure for the operator | During procedure
  Cumulative dose the operator receives as recorded from an electronic pocket dosimeter during the procedure.
Fluoroscopy Time | During procedure
  Total fluoroscopy utilized during the procedure as recorded by an Imaging System.
Safety event occurrence | From Day 0 to Day 3
  Medical device's safety event occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, Prof.MD, Principal Investigator — Het Ziekenhuisnetwerk Antwerpen vzw; Michael Haude, Prof.MD, Principal Investigator — Rheinland Klinikum Neuss GmbH
Locations (8):
- Het Ziekenhuisnetwerk Antwerpen vzw, Antwerp, Belgium
- France (3):
  - Brest university hospital, Brest, Brittany Region
  - Rouen university hospital, Rouen
  - Centre Cardiologique du Nord, Saint-Denis, Île-de-France Region
- Rheinland Klinikum Neuss GmbH, Neuss, Lukaskrankenhaus, Germany
- San Donato Policlinco Kardia, San Donato Milanese, MI, Italy
- Polskie Towarzystwo Kardiologiczne, Warsaw, Par Défaut, Poland
- Netcare Christiaan Barnard Memorial Hospital, Cape Town, le Cap, South Africa

IPD SHARING:
Plan to Share IPD: No